CLINICAL TRIAL: NCT02589652
Title: Efficacy of Switch or Sequential Combination Therapy of Pegylated Interferon Alfa-2a in Chronic Hepatitis B Patients With Low HBsAg and HBeAg Titers After Long-term Entecavir Therapy: A Multicenter, Prospective Cohort Study
Brief Title: Switch or Sequential Combination Therapy of Peginterferon in Hepatitis B Patients With Longterm Entecavir Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Other Study IDs: 81271833
Record Dates: First submitted 2015-10-25; First posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Hepatitis B
Keywords: Pegylated interferon; Entecavir
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a; entecavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Switch group: Patients who have been assigned to pegylated interferon alfa-2a.
  Interventions: Drug: Pegylated interferon alfa-2a
- Sequential combination group (S-C group): Patients who have been assigned to pegylated interferon alfa-2a plus entecavir.
  Interventions: Drug: Pegylated interferon alfa-2a plus Entecavir
- ETV group: Patients who have been assigned to entecavir monotherapy.
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Pegylated interferon alfa-2a — ETV 0.5mg oral daily plus PegIFN alfa-2a 180ug subcutaneous injection weekly for 8 weeks and followed by PegIFN alfa-2a 180ug subcutaneous injection weekly for 40 weeks
  Other Names: PegIFN alpha-2a
  Groups: Switch group
Drug: Pegylated interferon alfa-2a plus Entecavir — ETV 0.5mg oral daily plus PegIFN alfa-2a 180ug subcutaneous injection weekly for 48 weeks
  Other Names: PegIFN alpha-2a; ETV
  Groups: Sequential combination group (S-C group)
Drug: Entecavir — ETV 0.5mg oral daily for 48 weeks
  Other Names: ETV
  Groups: ETV group

SUMMARY:
This is a multicenter, prospective cohort study to evaluate the efficacy and safety of sequential combination or switch therapy of pegylated interferon alfa-2a in chronic hepatitis B patients with low HBsAg and HBeAg titers after long-term entecavir therapy, and compared to those who continued on ETV therapy.

DETAILED DESCRIPTION:
Chronic hepatitis B (CHB) infection remains a global health treat. The ideal end point of therapy is HBsAg loss or HBsAg seroconversion, indicating a complete remission of CHB. In patients with HBeAg-positive CHB, sustained HBeAg seroconversion is also a desirable end point. Current therapies include pegylated interferon (PegIFN) finite and nucleos(t)ide analogues (NUCs) longterm therapy. However, only 30-40% of patients may achieve HBeAg seroconversion on PegIFN monotherapy, whereas 15-20% of patients on entecavir (ETV). Recently, accumulating evidence had shown that optimization of switching or combining PegIFN in patients on long-term ETV therapy may increase rate of HBeAg seroconversion and even lead to the complete eradication of HBV. However, these two regimens has not been tested adequately in patients with low HBsAg/HBeAg titers on long-term ETV therapy.

This is a multicenter, prospective cohort study to evaluate the efficacy and safety of sequential combination or switch therapy of pegylated interferon alfa-2a in chronic hepatitis B patients with low HBsAg and HBeAg titers after long-term entecavir therapy, and compared to those who continued on ETV therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients > 18 and ≤ 60 years of age;
* Positive HBsAg for more than 6 months;
* Patients receiving previous ETV therapy ≥2 years;
* Patients who have achieved undetectable HBV DNA, HBsAg <1500IU/mL and HBeAg <200S/CO prior to switch or S-C therapy;
* ALT<=10*ULN and TB<2*ULN;
* Patients who have been assigned to treatment with PegIFN (S-C or switch) or continuous ETV after previous ETV therapy

Exclusion Criteria:

* Evidence of decompensated cirrhosis or hepatocellular carcinoma;
* Serological evidence of co-infection with HCV, HDV or HIV;
* Pregnant or breast-feeding women;
* Patients with diseases that might contraindicate to PegIFN therapy including severe psychiatric diseases, immunological diseases, severe retinopathy, thyroid dysfunction, leukocytopenia, thrombopenia, etc
* Patients receiving concomitant therapy with telbivudine;
* A history of drug or alcohol abuse;
* Other conditions that investigates consider not suitable for participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Chronic Hepatitis B Patients with Low HBsAg and HBeAg Titers after Long-term Entecavir Therapy
Sampling Method: Probability Sample
Enrollment: 294 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Rate of HBeAg seroconversion | week 72 (24 weeks after 48 weeks of treatment)
  Loss of HBeAg and detection of anti-HBe antibodies

SECONDARY OUTCOMES:
Rate of HBsAg loss | week 72 (24 weeks after 48 weeks of treatment)
  HBsAg loss with or without detection of anti-HBs antibodies
Rate of HBV DNA <20IU/mL | week 72 (24 weeks after 48 weeks of treatment)
Rate of HBsAg seroconversion | week 72 (24 weeks after 48 weeks of treatment)
Percentage of patients reaching a ≥ 1log10 decline of quantitative HBsAg | week 72 (24 weeks after 48 weeks of treatment)
Decline of quantitative HBsAg from baseline | week 72 (24 weeks after 48 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Zhang, MD, PhD, Principal Investigator — Huashan Hospital
Locations (17):
- China (17):
  - The First Affiliated Hospital, Anhui Medical University, Hefei, Anhui
  - The Second Affiliated Hospital, Anhui Medical University, Hefei, Anhui
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Fuzhou Municipal Infectious Disease Hospital, Fuzhou, Fujian
  - Zhongshan No.2 People's Hospital, Zhongshan, Guangdong, Guangzhou, Guangdong
  - The third People's Hospital of Shenzhen, Shenzhen, Guangdong
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Fifth People's Hospital of Suzhou, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - Shenyang Municipal Infectious Disease Hospital, Shenyang, Liaoning
  - Shandong Provincial Hospital of Shandong University, Jinan, Shandong
  - The First Affiliated Hospital Medical School of Xi'an Jiaotong University, Xi’an, Shanxi
  - The Affiliated Hospital of Luzhou Medical College, Luzhou, Sichuan
  - Sichuan Provincial People's Hospital, Sichuan, Sichuan
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The Second Hospital of Yinzhou of Ningbo, Ningbo, Zhejiang
  - Rui'an People's Hospital, Rui’an, Zhejiang